CLINICAL TRIAL: NCT00542802
Title: Multicenter, Comparative, Randomized, Open Trial to Evaluate Efficacy and Safety of Levetiracetam Versus Carbamazepine in Post Stroke Late Onset Crisis
Brief Title: Levetiracetam Versus Carbamazepine in Post-Stroke Late Onset Crisis
Acronym: EpIc
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scienze Neurologiche Ospedaliere (Other)
Responsible Party: Dr. Domenico Consoli, Scienze Neurologiche Ospedaliere
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EpIc 1151
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Epileptic Seizures; Stroke
Keywords: post stroke epileptic late onset seizures
MeSH Terms: conditions — Seizures; Stroke | interventions — Levetiracetam; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEV (Experimental): Levetiracetam
  Interventions: Drug: Levetiracetam
- CAR (Active Comparator): Carbamazepina
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam tablets 250-500 mg. The drug dosage will be up-titrated from 250 mg bid in the first 2 weeks to 500 mg bid during the rest of the treatment period. The dosage can be incremented until 1500 mg bid, at Investigator judgement if crisis continue, or it can be reduced in case of adverse events
  Arms: LEV
Drug: Carbamazepine — Carbamazepina tablets 200 mg. The drug dosage will be up-titrated from 100 mg die in the first 3 days to 100 mg bid during days 4 to 7, to 200 mg bid in the 2nd week, to 300 mg bid during the rest of the treatment period. The dosage can be incremented until 800 mg bid, at Investigator judgement if crisis continue, or it can be reduced in case of adverse events
  Arms: CAR

SUMMARY:
The principal purpose of the study is to determine the efficacy and safety of Levetiracetam versus Carbamazepine, intended as the number of patients free from crisis during the whole period of treatment, in patients affected by post stroke late onset crisis.

DETAILED DESCRIPTION:
Stroke is the most common cause of seizures in the elderly and seizures are among the most common sequelae of stroke.

About 10% of patients experience seizures since stroke onset up to several years (Silverman 2002). Arbitrarly a cut point of 2 weeks divide early seizures from late seizures (Honey 2000, Olofson 2000, Berger 1989).Late occurrence of late seizure appears to carry a high risk for epilepsy (Wilmore 1990).

The risk of epilepsy in some patients with a single stroke-related seizure is high enough to justify starting an anticonvulsant therapy before a second seizure occurs(Labovitz 2003).

Levetiracetam (S-α-ethil-2-oxo-pyrrolidine acetamide) is S-enantiomer of a pyrrolidine derivative and is unrelated to any other AED and has a unique preclinical and clinical profile (Gower et al 1992).

Levetiracetam (LEV) binds with a stereospecific binding site in the CNS that is saturable and reversible (Noyer 1995). This site actually known as LBS Levetiracetam Binding Site) is unique and do not correspond to any known receptor or channel that might be involved in neuroexcitability (Gillard 2003).

LEV selectively inhibits N-type Ca2 channels of CA1 pyramidal hyppocampal neurons (Lukyanetz et a 2002) and, despite of not having any activity on GABA-gated currents, it shows a potent ability to reverse the inhibitory effects of the negative allosteric modulators zinc and β-carbolines on both GABAA and glycine receptor mediated responses(Rigo et al. 2002).

LEV has no effects on normal neurons (Birnstiel et al.1997) LEV as other AEDs has effect in decreasing repetitive neuronal firing, but only LEV reduces the number of cells firing synchronously (amplitude) of the evoked PS(Margineau and Klitgaard 2000).

The efficacy profile of the drug has been established through three pivotal randomized double blind, placebo controlled, parallel studies on 904 patients suffering from partial seizures secondarily or not generalised that were not well controlled by previous treatment (Shorvon et al. 2000; Ben-Menachem et al. 2000; Cereghino et al. 2000).In these three studies LEV showed a significant reduction of seizure frequency. A pooled analysis of the results from these three studies supports a dose-response effect for levetiracetam: responder rates were 28.5, 34.3 and 41.3 % for patients treated with levetiracetam 1000, 2000, 3000 mg/day respectively, as compared with 13.1% for placebo group. The respective values for complete seizure freedom were 4.7, 6.3, 8.6 and 0.8%(Privitera 2002, Boon et al, 2002).

In a review of data for 1422 patients treated with levetiracetam, 38.6% of patients experienced a ≥ 50% reduction in seizure frequency and 20% experienced a reduction of ≥ 75%. The present study is not blinded because one of the purposes with the study has been to mimic daily clinical practice as close as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a stroke (ischemic and haemorrhagic) showing (one) subsequent seizure 14 days up to 3 years after stroke
* Patients has signed the informed consent form
* Aged ≥ 18 years

Exclusion Criteria:

* Severe stroke patients with Rankin scale > 3
* Patients with a life expectancy of < 12 months
* Patients screened more than 15 days after first seizure
* Patients with a diagnosed epilepsy
* Patients with clear evidence of myoclonic seizures
* Patients with contraindication to levetiracetam and carbamazepine use
* Patients presenting epileptic status at onset
* Patients having a MMSE <24
* Patients having a seizure before stroke
* Patients taking any AED 4 weeks prior to randomisation in the study
* Patients showing dysphagia after stroke not able to swallow tablets.
* Patients with a low compliance for the study
* Pregnant women, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method.
* Allergy or intolerance to pyrrolidine derivatives and/or tablet excipients or to carbamazepine derivates and /or tablet excipients
* Patients involved in another clinical trial 30 days prior randomization
* Patients with any tumour
* Patients with previous traumatic brain accident resulting in impairment of consciousness.
* Patients for whom it is not possible to assess seizure onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
number of patients free from post stroke recurrent crisis | one year

SECONDARY OUTCOMES:
To compare retention time of LEV vs CBZ since first intake throughout treatment period | one year
To compare time to second seizure in both treatments. | one year
To evaluate differences in cognitive function and in quality of life in levetiracetam and carbamazepine patients having post-stroke seizures at the end of treatment period | one year
evaluate EEG changes as compared with baseline with that obtained at the end of treatment period | one year
To compare seizure frequency in levetiracetam and carbamazepine groups throughout treatment period | one year
To evaluate the safety of levetiracetam versus carbamazepine throughout the treatment period | one year

CONTACTS AND LOCATIONS:
Overall Officials: domenico consoli, doctor, Principal Investigator — Ospedale Civile Vibo Valentia
Locations (24):
- Italy (24):
  - Ospedale S. Giacomo, Novi Ligure, AL
  - Ospedale S. Croce E Carle, Cuneo, CN
  - Ospedale S. Martino, Genova, GE
  - Istituto Clinico Humanitas, Rozzano, MI
  - USL 2 Ospedale B.G. Villa, Città della Pieve, PG
  - Ospedale Civile San Giovanni Battista di Foligno, Foligno, PG
  - Ospedale Santa Maria della Misericordia, Sant'Andrea Delle Fratte, PG
  - Istituto Neurologico C. Mondino, Pavia, PV
  - Ospedale Guzzardi, Vittoria, RG
  - Ospedale Di Portogruaro, Portogruaro, VE
  - Ospedale Civile, Vibo Valentia, VV
  - Policlinico Umberto I, Ancona
  - Ospedale A. Perrino, Brindisi
  - Ospedale Cannizzaro, Catania
  - Ospedale San Martino, Genova
  - Ospedale Civile Imperia ASL 1, Imperia
  - Ospedale A. Cardarelli-, Napoli
  - Ospedale Cardarelli, Napoli
  - Ospedale Civico, Palermo
  - Osp. Guglielmo da saliceto, Piacenza
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale SS. Annunziata - Ospedale Civile, Taranto
  - Ospedale Molinette-Università di Torino, Torino
  - Azienda Ospedaliera Universitaria Trieste, Trieste

REFERENCES:
- [Background] Silverman IE, Restrepo L, Mathews GC. Poststroke seizures. Arch Neurol. 2002 Feb;59(2):195-201. doi: 10.1001/archneur.59.2.195. PMID 11843689
- [Background] Stephen LJ, Brodie MJ. Epilepsy in elderly people. Lancet. 2000 Apr 22;355(9213):1441-6. doi: 10.1016/S0140-6736(00)02149-8. PMID 10791538
- [Background] Inzitari D. The Italian Guidelines for stroke prevention. The Stroke Prevention and Educational Awareness Diffusion (SPREAD) Collaboration. Neurol Sci. 2000 Feb;21(1):5-12. doi: 10.1007/s100720070112. No abstract available. PMID 10938196
- [Background] Hauser WA, Annegers JF, Kurland LT. Incidence of epilepsy and unprovoked seizures in Rochester, Minnesota: 1935-1984. Epilepsia. 1993 May-Jun;34(3):453-68. doi: 10.1111/j.1528-1157.1993.tb02586.x. PMID 8504780
- [Background] Bladin CF, Alexandrov AV, Bellavance A, Bornstein N, Chambers B, Cote R, Lebrun L, Pirisi A, Norris JW. Seizures after stroke: a prospective multicenter study. Arch Neurol. 2000 Nov;57(11):1617-22. doi: 10.1001/archneur.57.11.1617. PMID 11074794
- [Background] Rhoney DH, Tipps LB, Murry KR, Basham MC, Michael DB, Coplin WM. Anticonvulsant prophylaxis and timing of seizures after aneurysmal subarachnoid hemorrhage. Neurology. 2000 Jul 25;55(2):258-65. doi: 10.1212/wnl.55.2.258. PMID 10908901
- [Background] Olafsson E, Gudmundsson G, Hauser WA. Risk of epilepsy in long-term survivors of surgery for aneurysmal subarachnoid hemorrhage: a population-based study in Iceland. Epilepsia. 2000 Sep;41(9):1201-5. doi: 10.1111/j.1528-1157.2000.tb00326.x. PMID 10999560
- [Background] Berger AR, Lipton RB, Lesser ML, Lantos G, Portenoy RK. Early seizures following intracerebral hemorrhage: implications for therapy. Neurology. 1988 Sep;38(9):1363-5. doi: 10.1212/wnl.38.9.1363. PMID 3412583
- [Background] Sung CY, Chu NS. Epileptic seizures in thrombotic stroke. J Neurol. 1990 Jun;237(3):166-70. doi: 10.1007/BF00314589. PMID 2370564
- [Background] - Birnstiel S., Wulfert E., Beck SG., Levetiracetam (ucb L059) affects in vitro model of epilepsy in CA3 pyramidal neurons without altering normal synaptic transmission. Naunyn Schiemeberg Arch Pharmacol 1997: 356:611-618 - Bischoff U. And Schlobohm I. - Levetiracetam Has No Effect On Voltage-Gated Potassium Currents In Cultured Mouse Hippocampal Neurons. Epilepsia 43(Suppl. 8):88, 2002. - Blais L, Sheehy O, St-Hilaire JM, Bernier JP, Godfroid P, Le Lorier J. Economic evaluation of levetiracetam as adjunctive therapy in refractory epileptic patients. Value in Health 2002;5(6):509 - Boon P, Chauvel P, Pohlmann-Eden B, Otoul C, Wroe S. Dose-response effect of levetiracetam 1000 and 2000 mg/day in partial epilepsy. Epilepsy Research 2002;48:77-89
- [Background] - Castillo et al., Cochrane Database Syst Rev 2000;(3):CD 002028 - Chadwick et al., Cochrane Database Syst Rev 2002;(2):CD 001416 - Chaisewikul et al., Cochrane Database Syst Rev 2001;(1):CD 001901 - Coupez R., Nicolas JM, Browne TR Levetiracetam, a new antiepileptic agent: lack of in vitro and in vivo pharmacokinetic interaction with phenytoin in patient with valproic acid. Epilepsia 2003;44:171-178 - Cramer JA, Arrigo C, Van Hammee G, Gauer LJ, Cereghigno JJ. Effect of levetiracetam on epilepsy-related quality of life. Yhe N132 study group. Epilepsia 2000;41:868-874 - Cramer JA, Van Hammee G, N132 study Group. Maintenance of improvement in health-related quality of life during long-term treatment with levetiracetam. Epilepsy Behav 2003;4:118-123
- [Background] - Cramer J, De Rue K, Devinsky O, Edrich P, Trimble MR. A systematic review of the behavioral effects of levetiracetam in adults with epilepsy, cognitive disorder or an anxiety disorder during clinical trial. Epilepsy Behav. 2003;4:124-132 - Cramer JA, Ben-Menachem E, Franch J. Review of treatment options for refractory epilepsy: new medications and vagal nerve stimulation. Epilepsy Research 2001;47:17-25 - Cramer J.A., Leppik I.E., De Rue K., Eldrich P., Kramer G. - Tolerability of levetiracetam in elderly patients with CNS disorders - Epilepsy Research 2003; 56:135-145 - Devinsky O, Elger C. Efficacy of levetiracetam in partial seizure. Epileptic Disorder 2003;5(suppl 1):S27-S32
- [Background] - Ferrendelli J.A., French J., Leppik., Morrel M.J., Herbeuval A., Han J., Magnus L. - Use of levetiracetam in a population of patients aged 65 years and older: a subset analysis of the KEEPER trial - Epilepsy & Behavior 2003; 4:702-709 - French J, Edrich P, Cramer JA. A systematic review of safety profile of levetiracetam: a new antiepileptic drug. Epilepsy Res 2001;47:77-90 - Fucks B, Gillard M, Michel P, Lynch B, Vertongen P, Leprince P, Klitgaard H, Chatelain P. - Localisation and photoaffinity labelling of the levetriacetam dinding site in rat brain and certain cell lines Eur. J. Pharmacol 2003; 478, 11-19 - Gillard M, Fucks B, Michel P, Vertongen P, Massingham R, Chatelain P Binding characteristich of [3H]ucb 30889 to levetiracetam binding sites in rat brain Eur J Phamacol 2003; 478: 1-9
- [Background] - Giuliano RA, Hiersemenzel R, Baltes E, et al Influence of new antiepileptic drug (levetiracetam ucb L057) on the pharmacokinetics and pharmacodynamics of oral contraceptives Epilepsia 1996; 37 (Suppl.4):90 - Glauser TA, Pellock JM, Bebin EM. Efficacy and safety of levetiracetam in children with partial seizure: an open label trial. Epilepsia 2002;43:518-524 - Glauser TA, Dulac O. Preliminary efficacy of levetiracetam in children. Epileptic Disorder 2003;5(suppl 1):S45-S50 - Godfroid P, Hart Y, Roberts R, Le Lorier J. Seizure freedom in patients treated with adjunctive levetiracetam: economic evaluation within the NHS. Neurology 2003;60(S1):A433-A434 - Gower AJ, Hirsch E, Boehrer A, et al. Effects of levetiracetam, a novel antiepileptic drug on convulsant activity in two genetic rat models of epilepsy Epilepsy Research 1995; 22: 207-13
- [Background] - Gower AJ, Noyer M, Verloes R., et al. ucb L059, a novel anti-convulsant drug: pharmacological profle in animals. Eur J Pharmacol. 1992; 222: 193-203 - Gu J., Lynch B. A., Anderson D., Klitgaard H., Lu s., Elashoff M., Ebert U., Potschka H. - Loscher W. - The antiepileptic drug levetiracetam selectively modifies kindling-induced alterations in gene expression in the temporal lobe of rats. - European Journal of Neuroscience Vol. 19, pp334-345, 2004 - Kastelain-Nolst Trenitè DGA, Hirsch E. Levetiracetam: preliminary efficacy in generalised seizure. Epileptic Disorder 2003;5(suppl 1):S39-S44 - Klitgaard H, Matagne A, Gobert M, Michel P Evidence for a unique profile of levetiracetam in rodent models of seizures and epilepsy Eur. J. Pharmacology 1998; 353: 191-206
- [Background] - Klitgaard H, Pitkanen A, Antiepileptogenesis, neuroprotection, and disease modification in the treatment of epilepsy: focus on levetiracetam. Epileptic disorder 2003; 5:S9-S16 - Kraemer G, Eldrich P. Levetiracetam in Elderly patients with epilepsy - The American Eplepsy Society and The American Clinical Neurophysiology Society - Joint Meeting November 30-December 5, 2001 - Krakow K, Walker M, Otoul C, Sander JWAS. Long-term continuation of Levetiracetam in patients with refractory epilepsy. Neurology 2001;56:1772-1774 - Krauss GL, Abou-khalil B, Sheth SG. Efficacy of levetiracetam for treatment fo drug-resistant generalised epilepsy. Epilepsia 2001;42(suppl 7):181 - Krauss GL, Betts T, Abou-Khalil B, Bergey G, Yarrow H, Miller A. Levetiracetam treatment of idiopathic generalised epilepsy. Seizure 2003;12:617-620
- [Background] - Lagae L, Buyse G, Deconinck A, Ceulemans B. Effect of levetiracetam in refractory childhood epilepsy syndromes. Eur J Paediatric Neurol 2003;7:123-128 - Levy RH, Raguenau-Majlessi I, Baltes E Repeated administration of the novel antiepileptic agent levetiracetam does not alter digoxin pharmacokinetics and pharmacodynamics in healthy volunteers Epilepsy Research 2001; 47: 55-63 - Loscher W, Honak D, Rundfeld C Antiepileptogenic effect of the novel anticonvulsant levetiracetam (ucb L059) in the kindling model of temporal lobe epilepsy. - J. Pharmacological Exp. Ther 1998; 284: 474-9 - Lukyanetz EA, Shkryl VM, Kostyuk PG Selective blockade of N-type Calcium Channels by levetiracetam Epilepsia 2002; 43(1): 9-18 - Madeja M., Margineanu D.G., Gorji A., Siep E., Boerrigter P., Klitgaard H., Et Al.
- [Background] - Madeja M., Margineanu D.G., Gorji A., Siep E., Boerrigter P., Klitgaard H., Et Al. Reduction Of Voltage-Operated Potassium Currents By Levetiracetam: A Novel Antiepileptic Mechanism Of Action? - Neuropharmacology Oct-2003. 45(5):661-671. - Margineau D. G., Klitgaard Henrik Levetiracetam - Mechanism of action - Antiepilectic drugs, 5th edition. Edited by R.H. Levy, R.H. Mattson, B.S. Meldrum, and E.Perucca. Philadelphia: Lippincott Williams & Wilkins, 2002 - Margineau DG, Klitgaard H Inhibition of neural hyperynchrony in vitro differentiates levetiracetam fro classical antiepileptic drugs Pharmacol. Research 2000; 42(4): 281-285 - Marson AG, Hutton JL, Leach JP. Levetiracetam, Oxcarbazepine, Remacemide and zonisamide for drug resistant localization-related epilepsy: a systematic review. Epilepsy Res 2001;46:259-270
- [Background] - Marson AG, Kadir ZA, Hutton JL, Chadwick DW. The new antiepileptic drugs: a systematic review of their efficacy and tolerability. Epilepsia 1997;38:859-880 - Morrell MJ, Leppik I, French J, Ferrendelli J, Han J, Magnus L. The KEEPER trial: levetiracetam adjunctive treatment of partial-onset seizure in an open-label community-based study. Epilepsy Res 2003;54:153-161 - Niespodziany I, Klitgaard H, Margineau DG Desynchronizing effect of levetiracetam on epileptiform responses in rat hippocampal slices Neuropharmaology Neuroreport 2003; vol14(9): 1273-1276 - Noyer M, Gillard M, Magagne A., et al. The novel antiepileptic drug levetiracetam (ucb L059) appears o act via a specific binding site in CNS membranes. Eur J Pharmacol 1995 ; 286 : 137-146 - Patsalos PN Pharmacokinetic profile of levetiracetam: toward ideal characteristics. Pharmacol. Ther 2000; 83: 77-85 - Patsalos PN The pharmacokinetic characteristics of levetiracetam. Method Find. Exp. Clinic Pharmacol. 2003; 25: 123-129
- [Background] - Perucca E, Johannessen SI The ideal pharmacokinetic properties of an antiepileptic drug: how close does levetiracetam come? Epileptic Disorder 2003; 5(suppl 1):S17-S26 - Perucca E. Pharmacokinetics. In:Engel J Jr, Pedley TA Epilepsy-A comprehensive Textbook. New York: Raven Press 1997:1131-1153 - Radtke RA Pharmacokinetics of levetiracetam Epilepsia 2001; 42(Suppl 4):24-7 - Raguenau-Majlessi I, Levy RH, Meyerhoff C Lack of effect of repeated administration of levetiracetam on the pharmacodynamics and pharmakinetic profile of warfarin Epilepsy Res 2001; 47: 55-63 - Rigo JM, Hans G, Nguyen L, et al. The antiepileptic drug levetiracetam reverses the inhibition by negative allosteric modulators of neuronal GABA - and Glycine-gated current. Br J Pharmacol 2002; 136:659-72 - Sadek AH, Fix A, French J. Levetiracetam related behavioural adverse events: a post-marketing study. Epilepsia, 2002;43S8:151
- [Background] - Shorvon SD, Van Rijckevorsel. A new antiepileptic drug Levetiracetam, a pyrrolidone recently licensed as an antiepileptic drug. J Neurol Neurosurg Psychiatry 2002 ;72: 426-429 - Smith K, Betts T, Pritchett L. Levetiracetam, a promising option for the treatment of juvenile myoclonic epilepsy. Epilepsia 2000;41(suppl1):39 - Van Rijckevorsel K. The " number needed to treat " with levetiracetam : comparison with the other new antiepileptic drugs. Seizure 2001;10:235-236 - Welty TE, Gidal BE, Ficker DM, Privitera MD. Levetiracetam: a different approach to the pharmacotherapy of epilepsy. The Annals of Pharmacotherapy 2002;36:296-304 - Zona C, Niespodziany I, Marchetti C, et al. Levetiracetam does not modulate neuronal voltage-gated Na+ and T-type Ca2+ currents. Seizure 2001; 10: 279-86
- [Background] - Grigoletto Francesco, Zappalà Giuseppe, Anderson Dallas W., Lebowitz Barry D. Norms for the Mini.-Mental State Examination in a Healthy population. Neurology 1999;53:315-320 - Measso G., Zappalà G., Cavarzeran F, Crook TH, Romani L, Pirozzolo FJ, Grigoletto F., Amaducci LA, Lebowitz BD. Raven's colored progressive matrices: a normative study of a random sample of healthy adults. Acta Neurol. Scandinavica 1993:88:70-74 - Spinnler Hans & Tognoni Gianni Standardizzazione e taratura Italiana di Test Neuropsicologici Suppl. 8/to n.6 1987 The Italian Journal of Neurological Sciences - Zappalà G. Measso G., Cavarzeran F. Grigoletto F., Lebowitz B., Pirozzolo F., Amaducci L., Massari D., and Crook T. Aging and memory: corrections for age, sex and education fro three widely used memory tests - Italian Journal Of Neurological Sciences 1995;16: 177-184
- [Background] Ben-Menachem E, Falter U. Efficacy and tolerability of levetiracetam 3000 mg/d in patients with refractory partial seizures: a multicenter, double-blind, responder-selected study evaluating monotherapy. European Levetiracetam Study Group. Epilepsia. 2000 Oct;41(10):1276-83. doi: 10.1111/j.1528-1157.2000.tb04605.x. PMID 11051122
- [Background] Angehagen M, Margineanu DG, Ben-Menachem E, Ronnback L, Hansson E, Klitgaard H. Levetiracetam reduces caffeine-induced Ca2+ transients and epileptiform potentials in hippocampal neurons. Neuroreport. 2003 Mar 3;14(3):471-5. doi: 10.1097/00001756-200303030-00035. PMID 12634506
- [Background] - Arroyo S, Crawford P. Safety profile of levetiracetam. Epileptic Disorder 2003;5S1:S57-S63 - Ben-Menachem E, Edrich P, Van Vlyemen B, Sander JWAS, Schmidt B. Evidence for sustained efficacy of levetiracetam as add-on epilepsy therapy. Epilepsy Res 2003;53:57-64 - Ben-Menachem E. Preliminary efficacy of levetiracetam in monoterapy. Epileptic Disorder 2003;5(Suppl 1):S51-S55 - Betts T, Yarrow H, Greenhill L, Barrett M. Clinical experience of marketed levetiracetam in an epilepsy clinic - a one year follow-up study. Seizure 2003;12:140
- [Derived] Chang RS, Leung WC, Vassallo M, Sykes L, Battersby Wood E, Kwan J. Antiepileptic drugs for the primary and secondary prevention of seizures after stroke. Cochrane Database Syst Rev. 2022 Feb 7;2(2):CD005398. doi: 10.1002/14651858.CD005398.pub4. PMID 35129214